CLINICAL TRIAL: NCT02934750
Title: Effects of Pursed Lip Breathing on Exercise Capacity and Dyspnea in Patients With Interstitial Lung Disease: a Randomized Crossover Study
Brief Title: Pursed Lip Breathing in Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université du Québec a Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CE15.347
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-10

CONDITIONS: Interstitial Lung Disease
Keywords: pursed lip breathing; interstitial lund disease; exercise physiology
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pursed lip breathing (Experimental): In this arm, patients will be asked to perform a six-minute walking test while continuously using the pursed lip breathing technique.
  Interventions: Behavioral: Pursed lip breathing
- Usual breathing (No Intervention): In this control arm, patients will be asked to perform a six-minute walking test while breathing normally.

INTERVENTIONS:
Behavioral: Pursed lip breathing — Pursed lip breathing will be taught to the participants following the chronic obstructive pulmonary disease (COPD) Foundation recommendations:
  1. Breathe in through your nose (as if you are smelling something) for about 2 seconds.
  2. Pucker your lips like you're getting ready to blow out candles on a birthday cake.
  3. Breathe out very slowly through pursed-lips, two to three times as long as you breathed in.
  4. Repeat.
  Arms: Pursed lip breathing

SUMMARY:
This randomized, cross-over study aims at describing the effect of pursed lip breathing on exercise-induced dyspnea and exercise capacity in patients with interstitial lung disease.

DETAILED DESCRIPTION:
The use of pursed lip breathing (PLB) to improve exercise tolerance in COPD patients has been widely documented. However, its efficacy in patients with interstitial lung disease (ILD) has yet to be confirmed. This study aims to determine if PLB improves perceived exertion and exercise capacity during a six-minute walk test (6MWT) in patients with ILD. To achieve this, a prospective randomized crossover trial will be performed, in which patients with ILD and restrictive ventilatory defect will be recruited via the ILD clinic of Hôpital Notre-Dame. The study will be performed in a single visit, on the day where patients attend a routine physician-prescribed follow-up 6MWT. Patients will be asked to perform a total of two 6MWT. Patients will be randomized to perform the first test with or without using PLB, and the order will be reversed for the second test, with patients serving as their own control. During tests, ventilatory variables will be continuously measured using a portable metabolic cart. The observed parameters will be: perceived exertion using the Modified-Borg Scale, respiratory rate, minute-ventilation, heart rate, peripheral oxygen saturation, and 6-minute walk distance (6MWD). It is expected that the use of PLB will be associated with a decrease of at least one unit on the Modified Borg Scale, which would be clinically significant. Moreover, it is expected that the decrease in dyspnea with PLB will be related to a decrease in respiratory rate minute ventilation during 6MWT. The clinical impact of this study could be significant as therapies allowing the improvement of dyspnea in patients with ILD are scarce.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of interstitial lung disease, based on the results of a multidisciplinary diagnosis discussion.
* Restrictive ventilatory defect (i.e. total lung capacity (TLC) < 80% of predicted value) on pulmonary function testing.

Exclusion Criteria:

* Active cancer
* History of severe heart disease
* Neurological or orthopaedic problem that could interfere with exercise performance
* Physiological mixed syndromes (i.e. concomitant restrictive and obstructive defects)
* Exacerbation of disease or hospitalisation in the last 4 weeks prior to enrollment
* Long-term oxygen therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Exertional dyspnea | On the day of randomization
  Patient-reported dyspnea will be measured using the Borg scale

SECONDARY OUTCOMES:
Six-minute walking distance | On the day of randomization
Oxygen uptake (ml/min) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.
Carbon dioxide output (ml/min) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.
Respiratory rate (br/min) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.
Tidal volume (ml) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.
Minute-ventilation (l/min) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.
Peripheral oxygen saturation (%) | On the day of randomization, at each minute of the 6-minute walking test
  Non-invasive real-time measurements will be performed using a portable metabolic cart system.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno-Pierre Dubé, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal (CHUM)
Locations (1):
- CHUM (Notre-Dame Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parisien-La Salle S, Abel Rivest E, Boucher VG, Lalande-Gauthier M, Morisset J, Manganas H, Poirier C, Comtois AS, Dube BP. Effects of Pursed Lip Breathing on Exercise Capacity and Dyspnea in Patients With Interstitial Lung Disease: A RANDOMIZED, CROSSOVER STUDY. J Cardiopulm Rehabil Prev. 2019 Mar;39(2):112-117. doi: 10.1097/HCR.0000000000000387. PMID 30624373